CLINICAL TRIAL: NCT04821258
Title: Double-blind Randomized Clinical Trial to Evaluate the Effect of the Nutraceutical "MICODIGEST 2.0" on the Complications After Surgery With Curative Intent for Colorectal Cancer
Brief Title: Effect of the Nutraceutical "MICODIGEST 2.0" on the Complications After Surgery for Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: COGOMELO 2.0
Record Dates: First submitted 2021-03-23; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Cancer; Surgery--Complications
Keywords: Colorectal Cancer; Surgery Complications; Gut microbiota; Inflammatory pattern; Dietary pattern; Nutraceutical
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: CRC candidates for surgery with curative intent will be considered to include in the study. Patients who fulfill criteria will be screened and randomly allocated to be treated with MICODIGEST 2.0 or placebo previous to the admission. Patients will be also stratified based on tumor location (distal or proximal to splenic flexure).
  Patients will be followed for 4-6 weeks until surgery intervention.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MICODIGEST 2.0 supplement (Experimental): Treatment with MICODIGEST 2.0 will initiate with 10mL/day (before breakfast or before lunch) for 7 days, and rise to 20mL/day (10mL before breakfast and 10 mL before dinner) for 4-6 weeks.
  Interventions: Dietary Supplement: MICODIGEST 2.0 supplement
- Placebo (Placebo Comparator): Treatment with placebo will initiate with 10mL/day (before breakfast or before lunch) for 7 days, and rise to 20 mL/day (before breakfast and before dinner) for 4-6 weeks.
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: MICODIGEST 2.0 supplement — MICODIGEST is a nutraceutical which contains 9 different fungal extracts: Ganoderma lucidum, Agaricus blazei, Grifola frondosa, Hericium erinaceus, Cordyceps sinensis, Inonotus obliquus, Pleurotus ostreatus, Polyporus umbellatus y Lentinula edodes
  Arms: MICODIGEST 2.0 supplement
Dietary Supplement: Placebo supplement — Placebo
  Arms: Placebo

SUMMARY:
Most of Colorectal cancer (CRC) diagnosed are candidates for surgical resection with curative intent, although colorectal surgery is associated with some complications that could be life-threatening. Antibiotic prophylaxis is commonly used prior to the admission for the prevention of postoperative complications. However, this intervention can change the composition of intestinal microbiota and promote adverse inflammatory outcomes in CRC patients after surgery.

It seems the combination of different fungal extracts could be beneficial because of their role in gut microbiota modulation and their anti-inflammatory activity. Therefore, the fungal extract nutraceutical MICODIGEST 2.0 could be used to reduced the complications after CRC surgery.

Based on this hypothesis, we have designed a double-bind randomized clinical trial to evaluate the effect of MICODIGEST 2.0 on the complications after surgery with curative intent for CRC.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most common malignancies in western countries. Most of the CRC diagnosed are candidates for surgical resection with curative intent. Cure rates after surgery vary between 92 % and 67 % depending on the tumor stage. However, colorectal surgery is associated with some complications that could be life-threatening.

Antibiotic prophylaxis is commonly used prior to the admission for the prevention of this postoperative complications. Several studies have shown that antibiotic administration reduces the risk of infections associated with surgery. Nevertheless, this intervention does not modify the mortality and severity of other complications detected. Further, antibiotic prophylaxis could change the intestinal microbiota and promote adverse inflammatory outcomes in CRC patients after surgery.

Fungal polysaccharides have attracted attention because of their role in gut microbiota modulation. It seems that this type of polysaccharides could reduce pathogen levels and stimulate the growth of beneficial microorganism. Anti-inflammatory activity has also been described for these fungal polysaccharides. It seems the combination of different fungal extracts would send multiple stimuli to the immune system increasing intracellular reactions and interactions. Thus, the fungal extract nutraceutical MICODIGEST 2.0 could be used to reduced the complications after CRC surgery. MICODIGEST 2.0 is available since 2016 without any adverse effect reported.

For all these reasons we have designed a double-bind randomized clinical trial to evaluate the effect of MICODEGIST 2.0 on the complications after surgery with curative intent for CRC.

Apart from this purpose, we have also set the following secondary objectives:

* To evaluate the safety of MICODIGEST 2.0 in CRC patients.
* To evaluate the effect of MICODIGEST 2.0 on feal microbiome composition and diversity.
* To evaluate the effect of MICODIGEST 2.0 on inflammatory pattern, dietary pattern and quality of life.
* To analyze the effect of microbiome, inflammatory and dietary pattern on complications after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. CRC patients who are candidates for surgical treatment with curative intent (risk I-III).
2. American Society of Anesthesiologists' Physical Status Classification (ASA) <3.
3. Patients aged between 18 and 85 years.
4. Eastern Cooperative Oncology Group (ECOG) scale between 0-2.
5. Patients with preserved cognitive function.
6. Patient's authorization after reading the study information sheet.

Exclusion Criteria:

1. Candidates for neoadjuvant therapy.
2. Patients with concomitant carcinoma.
3. Allergy to the supplied nutraceutical or presence of malabsorption syndrome.
4. Presence of mental disorders
5. Patient with active infection or antibiotic therapy in the last month.
6. Previous colorectal surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Rate of complications. | week 4-6
  Anastomotic failure, infection, prolonged ileus, systemic complications and other will be measured. Clavien-Dindo classification will be used for grading the severity of these postoperative complications. These analysis will be measured to evaluate the effect of MICODEGIST 2.0 on the complications after surgery with curative intent for CRC.

SECONDARY OUTCOMES:
Frequency of adverse effects. | week 1-6
  Adverse effects will be considered during follow-up and after surgery using Common Terminology Criteria for Adverse Events (CTCAE) v5.0. This analysis will be measured to evaluate the safety of MICODIGEST 2.0 in CRC patients.
Fecal microbiome composition. | week 4-6
  High-quality DNA extraction will be performed in fecal samples. The bacterial 16S ribosomal ribonucleic acid gene will be sequencing on an Illumina MiSeq. Metagenomic species and a database with >200.000 strains will be used to define the microbiome composition. This analysis will be used to evaluate the effect of MICODIGEST 2.0 on feal microbiome composition.
Neutrophil/Lymphocyte ratio. | week 4-6
  Neutrophil/Lymphocyte will be measured dividing the absolute number of neutrophils by the absolute number of lymphocytes from peripheral blood sample. This inflammatory biomarker will be used to evaluate the effect of MICODIGEST 2.0 on inflammatory pattern.
C reactive protein (CRP) level. | week 4-6
  CRP levels (mg/dL) from peripheral blood samples will be measured to evaluate the effect of MICODIGEST 2.0 on inflammatory pattern.
Tumor Necrosis Factor alpha (TNF-alpha) and interleukin-6 (IL-6) levels. | week 4-6
  TNF-apha (pg/mL) and IL-6 (pg/mL) from peripheral blood samples will be measured to evaluate the effect of MICODIGEST 2.0 on inflammatory pattern.
Dietary pattern assessment. | week 4-6
  Patient-Generated Subjective Global Assessment survey (PG-SGA) will be used to assess the nutritional status. At the end of this survey, the patient will be rated nutritionally in one of three categories: "Well-nourished or anabolic" (PG-SGA - A), "Moderately or suspected of being undernourished" (PG-SGA B) and "Severely undernourished" (PG-SGA C). This analysis will be performed to evaluate the effect of MICODIGEST 2.0 on dietary pattern.
Quality of life assessment. | week 4-6
  The 36-item Short Form Health Survey (SF-36) will be used to measure the health-related quality-of-life. The SF-36 is a 36-item patient-reported questionnaire that covers eight health domains. Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state. This analysis will be perfomed to evaluate the effect of MICODIGEST 2.0 on quality of life.

REFERENCES:
- [Background] Gutierrez-Stampa MA, Aguilar V, Sarasqueta C, Cubiella J, Portillo I, Bujanda L. Impact of the faecal immunochemical test on colorectal cancer survival. BMC Cancer. 2020 Jul 1;20(1):616. doi: 10.1186/s12885-020-07074-y. PMID 32611328
- [Background] Gutierrez-Stampa MA, Aguilar V, Sarasqueta C, Cubiella J, Portillo I, Bujanda L. Colorectal Cancer Survival in 50- to 69-Year-Olds after Introducing the Faecal Immunochemical Test. Cancers (Basel). 2020 Aug 25;12(9):2412. doi: 10.3390/cancers12092412. PMID 32854370
- [Background] Cubiella J, Gonzalez A, Almazan R, Rodriguez-Camacho E, Fontenla Rodiles J, Dominguez Ferreiro C, Tejido Sandoval C, Sanchez Gomez C, de Vicente Bielza N, Lorenzo IP, Zubizarreta R. pT1 Colorectal Cancer Detected in a Colorectal Cancer Mass Screening Program: Treatment and Factors Associated with Residual and Extraluminal Disease. Cancers (Basel). 2020 Sep 6;12(9):2530. doi: 10.3390/cancers12092530. PMID 32899974
- [Background] Abis GSA, Stockmann HBAC, Bonjer HJ, van Veenendaal N, van Doorn-Schepens MLM, Budding AE, Wilschut JA, van Egmond M, Oosterling SJ; SELECT trial study group. Randomized clinical trial of selective decontamination of the digestive tract in elective colorectal cancer surgery (SELECT trial). Br J Surg. 2019 Mar;106(4):355-363. doi: 10.1002/bjs.11117. Epub 2019 Feb 25. PMID 30802304
- [Background] Espin Basany E, Solis-Pena A, Pellino G, Kreisler E, Fraccalvieri D, Muinelo-Lorenzo M, Maseda-Diaz O, Garcia-Gonzalez JM, Santamaria-Olabarrieta M, Codina-Cazador A, Biondo S. Preoperative oral antibiotics and surgical-site infections in colon surgery (ORALEV): a multicentre, single-blind, pragmatic, randomised controlled trial. Lancet Gastroenterol Hepatol. 2020 Aug;5(8):729-738. doi: 10.1016/S2468-1253(20)30075-3. Epub 2020 Apr 21. PMID 32325012
- [Background] Chowdhury AH, Adiamah A, Kushairi A, Varadhan KK, Krznaric Z, Kulkarni AD, Neal KR, Lobo DN. Perioperative Probiotics or Synbiotics in Adults Undergoing Elective Abdominal Surgery: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Ann Surg. 2020 Jun;271(6):1036-1047. doi: 10.1097/SLA.0000000000003581. PMID 31469748
- [Background] Tremaroli V, Backhed F. Functional interactions between the gut microbiota and host metabolism. Nature. 2012 Sep 13;489(7415):242-9. doi: 10.1038/nature11552. PMID 22972297
- [Background] Morowitz MJ, Babrowski T, Carlisle EM, Olivas A, Romanowski KS, Seal JB, Liu DC, Alverdy JC. The human microbiome and surgical disease. Ann Surg. 2011 Jun;253(6):1094-101. doi: 10.1097/SLA.0b013e31821175d7. PMID 21422915
- [Background] Ralls MW, Miyasaka E, Teitelbaum DH. Intestinal microbial diversity and perioperative complications. JPEN J Parenter Enteral Nutr. 2014 Mar-Apr;38(3):392-9. doi: 10.1177/0148607113486482. Epub 2013 May 1. PMID 23636012
- [Background] Ottosson F, Brunkwall L, Ericson U, Nilsson PM, Almgren P, Fernandez C, Melander O, Orho-Melander M. Connection Between BMI-Related Plasma Metabolite Profile and Gut Microbiota. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1491-1501. doi: 10.1210/jc.2017-02114. PMID 29409054
- [Background] Liu CJ, Zhang YL, Shang Y, Wu B, Yang E, Luo YY, Li XR. Intestinal bacteria detected in cancer and adjacent tissue from patients with colorectal cancer. Oncol Lett. 2019 Jan;17(1):1115-1127. doi: 10.3892/ol.2018.9714. Epub 2018 Nov 15. PMID 30655873
- [Background] Yin C, Noratto GD, Fan X, Chen Z, Yao F, Shi D, Gao H. The Impact of Mushroom Polysaccharides on Gut Microbiota and Its Beneficial Effects to Host: A Review. Carbohydr Polym. 2020 Dec 15;250:116942. doi: 10.1016/j.carbpol.2020.116942. Epub 2020 Aug 27. PMID 33049854
- [Background] Ma G, Kimatu BM, Zhao L, Yang W, Pei F, Hu Q. In vivo fermentation of a Pleurotus eryngii polysaccharide and its effects on fecal microbiota composition and immune response. Food Funct. 2017 May 24;8(5):1810-1821. doi: 10.1039/c7fo00341b. PMID 28513745
- [Background] Chang CJ, Lin CS, Lu CC, Martel J, Ko YF, Ojcius DM, Tseng SF, Wu TR, Chen YY, Young JD, Lai HC. Ganoderma lucidum reduces obesity in mice by modulating the composition of the gut microbiota. Nat Commun. 2015 Jun 23;6:7489. doi: 10.1038/ncomms8489. PMID 26102296
- [Background] Diling C, Chaoqun Z, Jian Y, Jian L, Jiyan S, Yizhen X, Guoxiao L. Immunomodulatory Activities of a Fungal Protein Extracted from Hericium erinaceus through Regulating the Gut Microbiota. Front Immunol. 2017 Jun 12;8:666. doi: 10.3389/fimmu.2017.00666. eCollection 2017. PMID 28713364
- [Background] Nowak R, Nowacka-Jechalke N, Juda M, Malm A. The preliminary study of prebiotic potential of Polish wild mushroom polysaccharides: the stimulation effect on Lactobacillus strains growth. Eur J Nutr. 2018 Jun;57(4):1511-1521. doi: 10.1007/s00394-017-1436-9. Epub 2017 Mar 28. PMID 28353071
- [Background] Hess J, Wang Q, Gould T, Slavin J. Impact of Agaricus bisporus Mushroom Consumption on Gut Health Markers in Healthy Adults. Nutrients. 2018 Oct 2;10(10):1402. doi: 10.3390/nu10101402. PMID 30279332
- [Background] Barbieri A, Quagliariello V, Del Vecchio V, Falco M, Luciano A, Amruthraj NJ, Nasti G, Ottaiano A, Berretta M, Iaffaioli RV, Arra C. Anticancer and Anti-Inflammatory Properties of Ganoderma lucidum Extract Effects on Melanoma and Triple-Negative Breast Cancer Treatment. Nutrients. 2017 Feb 28;9(3):210. doi: 10.3390/nu9030210. PMID 28264501
- [Background] Chen X, Hu ZP, Yang XX, Huang M, Gao Y, Tang W, Chan SY, Dai X, Ye J, Ho PC, Duan W, Yang HY, Zhu YZ, Zhou SF. Monitoring of immune responses to a herbal immuno-modulator in patients with advanced colorectal cancer. Int Immunopharmacol. 2006 Mar;6(3):499-508. doi: 10.1016/j.intimp.2005.08.026. Epub 2005 Sep 15. PMID 16428086
- [Background] Nie Y, Lin Q, Luo F. Effects of Non-Starch Polysaccharides on Inflammatory Bowel Disease. Int J Mol Sci. 2017 Jun 27;18(7):1372. doi: 10.3390/ijms18071372. PMID 28654020
- [Background] Jiang J, Wojnowski R, Jedinak A, Sliva D. Suppression of proliferation and invasive behavior of human metastatic breast cancer cells by dietary supplement BreastDefend. Integr Cancer Ther. 2011 Jun;10(2):192-200. doi: 10.1177/1534735410386953. Epub 2010 Oct 6. PMID 20926736
- [Background] Jakopovich I. New dietary supplements from medicinal mushrooms: Dr Myko San--a registration report. Int J Med Mushrooms. 2011;13(3):307-13. doi: 10.1615/intjmedmushr.v13.i3.110. PMID 22135883
- [Background] Rai SN, Mishra D, Singh P, Vamanu E, Singh MP. Therapeutic applications of mushrooms and their biomolecules along with a glimpse of in silico approach in neurodegenerative diseases. Biomed Pharmacother. 2021 May;137:111377. doi: 10.1016/j.biopha.2021.111377. Epub 2021 Feb 15. PMID 33601145
- [Background] Borchers AT, Krishnamurthy A, Keen CL, Meyers FJ, Gershwin ME. The immunobiology of mushrooms. Exp Biol Med (Maywood). 2008 Mar;233(3):259-76. doi: 10.3181/0708-MR-227. PMID 18296732
- [Background] Wasser SP. Current findings, future trends, and unsolved problems in studies of medicinal mushrooms. Appl Microbiol Biotechnol. 2011 Mar;89(5):1323-32. doi: 10.1007/s00253-010-3067-4. Epub 2010 Dec 29. PMID 21190105
- [Derived] Regueiro C, Codesido L, Garcia-Nimo L, Zarraquinos S, Remedios D, Rodriguez-Blanco A, Sinde E, Fernandez-de-Ana C, Cubiella J. Effect of the Nutraceutical Micodigest 2.0 on the Complication Rate of Colorectal Cancer Surgery With Curative Intent: Protocol for a Placebo-Controlled Double-blind Randomized Clinical Trial. JMIR Res Protoc. 2022 May 16;11(5):e34292. doi: 10.2196/34292. PMID 35576566
- See also: World Health Organization. Cancer Today. International Agency for Research on Cancer. (2020) — https://gco.iarc.fr/today/home